CLINICAL TRIAL: NCT04669210
Title: A Randomized, Multicenter, Open-label Phase II Trial to Compare Prophylaxis of Graft Versus Host Disease With Tacrolimus and Mycophenolate Mofetil Versus Ruxolitinib After Post-transplant Cyclophosphamide
Brief Title: PTCy and Ruxolitinib vs PTCy, Tacrolimus and MMF in MUD and Haploidentical HSCT
Acronym: PTCyRuxo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, Ivan S Moiseev, RM Gorbacheva Research institute scientific director, St. Petersburg State Pavlov Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CINC424ARU01T
Record Dates: First submitted 2020-11-26; First posted 2020-12-16 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Graft-versus-host-disease; Stem Cell Transplant Complications; Acute Myeloid Leukemia; Acute Lymphoid Leukemia
Keywords: Graft-versus-host-disease; Prophylaxis; ruxolitinib; tacrolimus; MMF; PTCY; cyclophosphamide; unrelated donor; haploidentical donor; randomized trial
MeSH Terms: conditions — Graft vs Host Disease; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — ruxolitinib; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PTCY tacrolimus MMF (Active Comparator): Conditioning:
  fludarabine 180 mg/m2 busulfan 8-14 mg/kg per os
  GVHD prophylaxis:
  cyclophosphamide 50 mg/kg day+3, +4 tacrolimus 0.03 mg/kg from day+5 to 100 mycophenolate mofetil 30 mg/kg from day+5 to 35
  Interventions: Drug: Tacrolimus; Drug: Mycophenolate Mofetil
- PTCY ruxolitinib (Experimental): Conditioning:
  fludarabine 180 mg/m2 busulfan 8-14 mg/kg per os ruxolitinib 5 mg tid days -7 to -2
  GVHD prophylaxis:
  cyclophosphamide 50 mg/kg day+3, +4 ruxolitinib 5 mg tid days +5 to +21 ruxolitinib 5 mg bid days +22 to +150
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib administered during conditioning 5 mg tid before allogeneic hematopoietic stem cell transplantation, 5 mg tid days 5-21 and 5 mg bid days 22-150 after transplantation instead of tacrolimus and MMF.
  Other Names: Jakavi
  Arms: PTCY ruxolitinib
Drug: Tacrolimus — Tacrolimus 0.03 mg/kg adjusted to concentrations 5-15 ng/ml from day+5 to +100
  Other Names: Prograf
  Arms: PTCY tacrolimus MMF
Drug: Mycophenolate Mofetil — Mycophenolate mofetil 30 mg/kg from day +5 to +35
  Other Names: CellCept
  Arms: PTCY tacrolimus MMF

SUMMARY:
This is multicenter investigator-initiated randomized open-label phase II clinical trial to compare prophylaxis of graft versus host disease treated with tacrolimus and mycophenolate mofetil versus ruxolitinib after post-transplant cyclophosphamide.

In total 128 patients will be included in the study. After inclusion into the study and performing of transplantation patients will be randomized in 1:1 proportion in two arms (64 patients per arm): arm A will include patients who will be treated with cyclophosphamide and ruxolitinib for GVHD prophylaxis; arm B will include patients who will be treated with cyclophosphamide, tacrolimus and MMF for GVHD prophylaxis. After the end of the treatment patients will be followed-up during two years.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent to participate in the study, signed by the patient;
2. Diagnosis: acute lymphoblastic or acute myeloblastic leukemia;
3. Morphological remission, defined as less than 5% of blasts by microscopy or flow cytometry with a peripheral leukocyte level of more than 1.500 μL. It is acceptable to include patients without restored platelets or erythrocytes;
4. Indications for performing allogeneic hematopoietic stem cell transplantation, determined by the participating center in accordance with local medical practice;
5. Unrelated or haploidentical donor;
6. Age 18-70 years;
7. Functional status according to ECOG scale 0-2 score.

Exclusion Criteria:

1. Repeated allogeneic transplantation, regardless of the indications for its implementation;
2. Source of graft - umbilical cord stem cells;
3. Any ex vivo modification of the graft with the exception of separation or washing of red blood cells;
4. The presence of more than 5% of clonal tumor cells according to flow cytometry in the presence of morphological remission;
5. Diagnosis: acute promyelocytic leukemia;
6. Severe organ failure: creatinine more than 2 ULN; ALT, AST more than 5 ULN; bilirubin more than 1.5 ULN; respiratory failure more than 1 grade;
7. Unstable hemodynamics, requiring the introduction of vasopressors;
8. Uncontrolled bacterial or fungal infection at the time of randomization, determined by the level of CRP> 70 mg/l with adequate antibacterial or antifungal therapy;
9. Rhythm disturbances that persist despite adequate antiarrhythmic therapy: a tachysystolic form of atrial fibrillation, ventricular arrhythmias V gradation according to Laun, AV block of III degree;
10. Decrease in ejection fraction according to echocardiography less than 40%;
11. Angina of more than II functional class or unstable angina;
12. Another severe concomitant pathology, which according to the attending physician does not allow the patient to be included in the study;
13. Pulmonary pathology with a decrease in FEV1 of less than 60% or pulmonary diffusion capacity of less than 60%;
14. Inability to quit smoking for up to 6 months after transplantation;
15. Pregnancy or refusal to perform highly effective contraception for 6 months after transplantation.

    Highly effective contraceptive methods include:
    * Total abstinence: if it corresponds to the preferred and customary way of life of the patient. Periodic abstinence (for example, calendar, ovulation, symptothermal, postovulation methods) and interrupted sexual intercourse are not considered acceptable methods of contraception;
    * Female sterilization (surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy or tubal ligation at least 6 weeks before the start of the therapy being studied. In the case of ovariectomy only, the reproductive status of the woman must be confirmed using a subsequent analysis of hormones;
    * Sterilization of the male partner (at least 6 months before screening). For women participating in the study, the sexual partner after a vasectomy should be the only partner;
    * Use of oral, injectable or implanted hormonal contraceptive drugs, intrauterine devices or contraceptive systems, or other forms of hormonal contraception with similar efficacy (failure rate less than 1%), for example, hormonal vaginal rings or transdermal hormonal contraceptives.
16. Somatic or mental pathology not allowing to sign informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Incidence of acute GVHD grade II-IV | 125 days
  Proportion of patients with acute GVHD II-IV grade

SECONDARY OUTCOMES:
Non-relapse mortality | 2 years
  Cumulative incidence of patients with mortality without hematological relapse of malignancy
Relapse incidence | 2 years
  Cumulative incidence of patients with relapse
Incidence of moderate and severe chronic GVHD | 2 years
  Cumulative incidence of patients with moderate and severe chronic GVHD according to NIH 2015 criteria
Overall survival | 2 years
  Kaplan-Meier estimate of death from all causes
Event-free survival | 2 years
  Kaplan-Meier estimate of death or relapse
Incidence of HSCT-associated adverse events (safety and toxicity) | 125 days
  Toxicity assessment is based on NCI CTC AE 5.0 grades. Veno-occlusive disease incidence and severity assessment is based on EBMT criteria 2016. Transplant-associated microangiopathy incidence assessment is based on Cho et al. criteria. All toxicity measurements will be aggregated as severity scores.
Primary or secondary graft failure | 2 years
  Cumulative incidence of patients with primary or secondary graft failure defined by the absence of donor chimerism.
Incidence of infections | 6 months
  Number of patients with bacteremia before engraftment, bacteremia after engraftment, severe sepsis (presence of multiple organ failure), pneumonia, soft tissue infection, invasive mycosis (probable or proven invasive aspergillosis, candidaemia, zygomycosis), reactivation of cytomegalovirus, other opportunistic viral infections

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - National Hematology Research Center, Moscow
  - RM Gorbacheva Research Institute, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Access Criteria: Per request to the Ethical Committee of Pavlov University with the study plan and rationale for the use of the data.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/10/NCT04669210/Prot_SAP_000.pdf